CLINICAL TRIAL: NCT03495141
Title: Simbionix GI Mentor Simulated Endoscopy Training
Brief Title: Outcomes in Simulated Endoscopy Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 8244
Record Dates: First submitted 2018-03-13; First posted 2018-04-11 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Impact of Supervision on Endoscopy Simulation Curriculum
MeSH Terms: interventions — Organization and Administration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will not know who was randomized to supervised versus unsupervised simulator training.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised (Active Comparator): Participants first take part in supervised/coached colonoscopy module session twice (case one and case two) and then transition to performing an unassisted colonoscopy module twice (case three and case four).
  Interventions: Behavioral: Supervision/Coaching
- Unsupervised (Active Comparator): Participants will either first partake in an unsupervised colonoscopy module twice (case one and case two) and then transition to a supervised/coached colonoscopy module session twice (case three and case four).
  Interventions: Behavioral: Supervision/Coaching

INTERVENTIONS:
Behavioral: Supervision/Coaching — Supervision involves coaching the trainee on insertion and withdrawal technique in a standard colonoscopy in a novice trainee

SUMMARY:
Eligible participants are those who are members of the general surgery residency pediatric gastroenterology fellowship, and adult gastroenterology fellowship. Through a randomized-controlled trial, participants will fill out a baseline set of demographic information including year of training, approximate number of colonoscopies to date, specialty, age, sex and handedness. Participation in this activity is completely voluntary. Trainees will be randomized to one of two groups. Either first participating in an unassisted colonoscopy module twice and then taking a questionnaire and then transitioning to a supervised/coached colonoscopy module session twice and taking a questionnaire, versus the reverse, in which the participant first partakes in a supervised/coached colonoscopy module session twice and then transitions to performing a colonoscopy module twice, unassisted. Objective measures will be assessed by the module software and supervising faculty. Specifically, using individuals' survey responses to see if early supervision improves survey scores. Survey questions focus on student learning, completing module objectives and faculty performance in simulation. The survey will also ask subjects to self-rate their scores and comfort level with endoscopy skills. Survey responses will not be linked to an individuals' performance in their program training and endoscopy coaches will not be made aware of the survey responses.

DETAILED DESCRIPTION:
This will be a randomized controlled trial in which eligible participants will be members of the general surgery residency and adult gastroenterology fellowship. Investigators will ask all consenting participants to fill out a baseline set of demographic information including their year of training, the approximate number of colonoscopies to date, specialty, age, sex and dominant-handedness. Additional questions to be asked will inquire about the participant's experience in regard to the unassisted and supervision/coached colonoscopy module experience. Participation in this activity is completely voluntary, and the participating trainee is under no obligation to complete or finish the simulation or subsequent surveys The participant will be randomized to one of two groups. A computer program will make this random assignment. Neither the participant nor their physician coach will be able to choose which group they will be in. Participants will either first partake in an unassisted colonoscopy module twice (case one and case two) and then transition to a supervised/coached colonoscopy module session twice (case three and case four). The alternative is in which the participant first partakes in a supervised/coached colonoscopy module session twice (case one and case two) and then transitions to performing an unassisted colonoscopy module twice (case three and case four). A questionnaire examining training experience will be administered after case # 4 in both groups. This survey will take approximately 5 minutes to complete. Other objective measures will be assessed by supervising faculty and other metrics acquired through the simulator software. Individuals' survey responses will be used to see if early supervision improves trainee satisfaction and perceptions on survey scores. Participants will attend one individual training session date that will satisfy the designed simulation experience. The trainee can stop participating in this study at any time and participation in the study is voluntary and trainees may choose not to participate. It is important to note that refusal to participate will not affect a learner's access to the training center and will not affect their standing in their respective training program. The results will not be included in their official training record. Note no prior procedural or technical knowledge is required. Enrollment will continue for the 2018-2019 academic year and possibly academic years thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Consenting trainees of adult and pediatric gastroenterology fellowships and general surgery residencies at the University of Oklahoma Health Sciences Center.

Exclusion Criteria:

* Unwilling to consent.

Ages: 22 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-03-06 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of mucosa inspected | through study completion, an average of 1 year
  The primary outcome will be the difference in percentage of mucosa inspected between the two study groups based on the report of the simulator after each of 4 predefined cases

SECONDARY OUTCOMES:
Time to reach cecum | through study completion, an average of 1 year
  Time to reach cecum after time of colonoscope insertion
Participant satisfaction score | through study completion, an average of 1 year
  Participants will be asked to self-report satisfaction with supervised and unsupervised endoscopic simulator experiences

CONTACTS AND LOCATIONS:
Overall Officials: William Tierney, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No
Participant data will only be known to PI and co-investigator (this writer) and de-identified data will be used for statistical analysis.